CLINICAL TRIAL: NCT00001196
Title: Evaluation of Salivary Gland Dysfunction
Status: Terminated | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 840056; 84-D-0056
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-09-29

CONDITIONS: Sjogren's Syndrome; Salivary Gland
Keywords: Salivary Function; Salivary Gland; Sjogren's Syndrome; Dry Mouth
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will evaluate patients with complaints of dry mouth to determine the cause and severity of their salivary gland dysfunction and their possible eligibility for other NIDCR protocols. Salivary gland secretions have antibacterial, lubricatory, remineralizing, digestive, buffering and cleansing properties. Impaired function of these glands can cause an increase in tooth decay; a variety of oral hard and soft tissue changes, with painful, burning, or ulcerated oral mucosal; problems chewing, swallowing, and speaking; and diminished taste and smell.

Patients with dry mouth complaints suggestive of salivary gland dysfunction may be eligible for this study. In addition, patients with recent onset of arthritis may enroll. Patients with arthritis are at risk for developing a disorder called Sjogren's syndrome, in which the glands that produce saliva may be damaged.

Participants will have a complete medical and dental history. Saliva samples will be collected from the major salivary glands, which are located in the cheeks and under the jaw. Several blood samples will also be drawn for tests. Some patients will have a biopsy of the minor salivary glands, usually from the lower lip, to confirm or rule out the diagnosis of Sjogren's syndrome and determine the extent of changes in the salivary glands. The ability to taste and smell may also be evaluated, and patients may have an ultrasound examination of their swallowing function.

DETAILED DESCRIPTION:
This study will evaluate participants with complaints of dry mouth to determine the cause and severity of their salivary gland dysfunction and their possible eligibility for other NIDCR protocols. Salivary secretions have antibacterial, lubricating, remineralizing, digestive, buffering and cleansing properties. Impaired function of these glands can cause an increase in tooth decay; a variety of oral hard and soft tissue changes, with painful, burning or ulcerated or oral mucosa; problems chewing, swallowing and speaking; and diminished taste and smell.

Participants with dry mouth complaints suggestive of salivary gland dysfunction may be eligible for this study.

Participants will have a complete medical and dental history. Saliva samples will be collected from the major salivary glands, which are located in the cheeks and under the tongue. Several blood samples will also be drawn for tests. Some participants will have a biopsy of the minor salivary glands, usually from inside the lower lip, to confirm or rule out the diagnosis of Sj(SqrRoot)(Delta)gren s syndrome and to determine the extent of changes in the salivary glands. An eye examination including a standard eye examination and a dry eye assessment is done. The ability to taste and smell may also be evaluated, and participants may have an ultrasound examination of their swallowing function.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must have dry mouth symptoms (xerostomia) or a reasonable clinical suspicion of having Sj(SqrRoot)(Delta)gren s syndrome or other salivary gland disease
  2. Ability to provide informed consent.

EXCLUSION CRITERIA:

a. Age less than 12 years.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1740 (Actual)
Dates: Start 1984-03-23; Study Completion 2015-09-29

PRIMARY OUTCOMES:
To determine the cause and severity of the subject's saivary gland dysfunction. | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Ilias G Alevizos, D.M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fox PC, van der Ven PF, Sonies BC, Weiffenbach JM, Baum BJ. Xerostomia: evaluation of a symptom with increasing significance. J Am Dent Assoc. 1985 Apr;110(4):519-25. doi: 10.14219/jada.archive.1985.0384. PMID 3858368
- [Background] Daniels TE, Fox PC. Salivary and oral components of Sjogren's syndrome. Rheum Dis Clin North Am. 1992 Aug;18(3):571-89. PMID 1496162
- [Background] Fox PC, Speight PM. Current concepts of autoimmune exocrinopathy: immunologic mechanisms in the salivary pathology of Sjogren's syndrome. Crit Rev Oral Biol Med. 1996;7(2):144-58. doi: 10.1177/10454411960070020301. PMID 8875029
- [Derived] Tanaka T, Warner BM, Odani T, Ji Y, Mo YQ, Nakamura H, Jang SI, Yin H, Michael DG, Hirata N, Suizu F, Ishigaki S, Oliveira FR, Motta ACF, Ribeiro-Silva A, Rocha EM, Atsumi T, Noguchi M, Chiorini JA. LAMP3 induces apoptosis and autoantigen release in Sjogren's syndrome patients. Sci Rep. 2020 Sep 16;10(1):15169. doi: 10.1038/s41598-020-71669-5. PMID 32939030
- [Derived] Burbelo PD, Ferre EMN, Chaturvedi A, Chiorini JA, Alevizos I, Lionakis MS, Warner BM. Profiling Autoantibodies against Salivary Proteins in Sicca Conditions. J Dent Res. 2019 Jul;98(7):772-778. doi: 10.1177/0022034519850564. Epub 2019 May 16. PMID 31095438
- [Derived] Alevizos I, Alexander S, Turner RJ, Illei GG. MicroRNA expression profiles as biomarkers of minor salivary gland inflammation and dysfunction in Sjogren's syndrome. Arthritis Rheum. 2011 Feb;63(2):535-44. doi: 10.1002/art.30131. PMID 21280008